CLINICAL TRIAL: NCT00147290
Title: ADVANCE CRT - D: ATP Delivery for Painless ICD Therapy
Brief Title: ADVANCE CRT - D: Antitachycardia Pacing (ATP) Delivery for Painless Implantable Cardioverter Defibrillator (ICD) Therapy
Acronym: ADVANCE-CRTD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Elisabetta Santi, Medtronic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 400ACRT
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2015-08

CONDITIONS: Tachycardia, Ventricular; Ventricular Fibrillation
Keywords: ATP; Tachycardia; CRT-D
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Tachycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BiV (Experimental): ATP therapies are delivered in both the ventricles
  Interventions: Device: Implantable Cardiac Defibrillator
- RV (Active Comparator): ATP delivered only in the right ventricle
  Interventions: Device: Implantable Cardiac Defibrillator

INTERVENTIONS:
Device: Implantable Cardiac Defibrillator — Implantable cardiac defibrillator with programmable Fast Ventricular tachycardia detection (FVT) window
  Other Names: ICD

SUMMARY:
To compare the efficacy of RV and BiV ATP for the termination of ventricular arrhythmias in patients who are candidates to a cardiac resynchronisation therapy (CRT) and have a Class I or IIA indication for ICD implantation.

The hypothesis of delivering ATP from different sites (RV or BIV) has never been evaluated in a prospective, controlled and randomized study.

DETAILED DESCRIPTION:
Main objective: Compare efficacy of ATP therapy (Burst, 8 pulses, 88 %, 1 sequence) to terminate all types of ventricular tachycardia (all VTs (FVT+VT)) when delivered in the right ventricle (RV) only versus both ventricles (BiV) resulting in a 10 % difference in favour of BIV ATP

Secondary objectives:

* Compare efficacy of the first BiV and RV ATP (Burst, 8 pulses, 88 %) to terminate fast ventricular tachycardia (FVT)
* Compare efficacy of the first BiV and RV ATP (Burst, 8 pulses, 88 %) to terminate slow ventricular tachycardia (slow VT)
* Compare efficacy of BiV and RV ATP (all ATP therapies) to terminate slow ventricular tachycardia (slow VT)
* Determine the rate of both FVT and VT episodes which are accelerated or degenerates into VF

ELIGIBILITY:
Inclusion Criteria:

* CRT + ICD indications (Class I-IIA) according to the guidelines
* Patients have been implanted with a Medtronic Marquis Family ICD capable of RV-ATP or BIV-ATP
* Patients in chronic AF who undergo a complete AV ablation and that the complete AV block is confirmed at PHD

Exclusion Criteria:

* Patient's life expectancy less than 1 year due to a non cardiac chronic disease
* Patient on heart transplant list which is expected in < 1 year
* Patient's age less than 18 years
* Replacements and upgrades
* Epicardial lead
* Mechanical tricuspid valve
* Ventricular Tachyarrhythmias associated with reversible causes
* Unwillingness or inability to provide written informed consent
* Enrollment in, or intention to participate in, another clinical study during the course of this study
* Inaccessibility for follow-up at the study center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2004-02; Primary Completion 2007-04 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Gasparini, Dr., Principal Investigator — Istituto Clinico Humanitas Mirasole SpA; Mario Bocchiardo, Dr., Principal Investigator — Ospedale Civile di Asti; Antonio Curnis, Dr., Principal Investigator — Spedali Civili di Brescia; Rafael Peinado, Dr., Principal Investigator — La Paz Madrid; Philippe Mabo, Prof., Principal Investigator — Rennes University Hospital; Thomas Lavergne, Dr., Principal Investigator — E. H. Pompidou - Paris; Frederic Anselme, Dr., Principal Investigator — University Hospital, Rouen; Joerg Schwab, Dr., Principal Investigator — University Clinic - Bonn
Locations (1):
- Medtronic Italia SpA, Sesto San Giovanni, Milan, Italy

REFERENCES:
- [Background] Schwab JO, Gasparini M, Anselme F, Mabo P, Peinado R, Lavergne T, Bocchiardo M, Mascioli G, Passardi M, Mainardis M. Right ventricular versus biventricular antitachycardia pacing in the termination of ventricular tachyarrhythmia in patients receiving cardiac resynchronization therapy: the ADVANCE CRT-D trial. J Cardiovasc Electrophysiol. 2006 May;17(5):504-7. doi: 10.1111/j.1540-8167.2006.00433.x. PMID 16684023
- [Derived] Landolina M, Boriani G, Biffi M, Cattafi G, Capucci A, Dello Russo A, Facchin D, Rordorf R, Sagone A, Del Greco M, Morani G, Nicolis D, Meloni S, Grammatico A, Gasparini M. Determinants of worse prognosis in patients with cardiac resynchronization therapy defibrillators. Are ventricular arrhythmias an adjunctive risk factor? J Cardiovasc Med (Hagerstown). 2022 Jan 1;23(1):42-48. doi: 10.2459/JCM.0000000000001236. PMID 34392257
- [Derived] Gasparini M, Kloppe A, Lunati M, Anselme F, Landolina M, Martinez-Ferrer JB, Proclemer A, Morani G, Biffi M, Ricci R, Rordorf R, Mangoni L, Manotta L, Grammatico A, Leyva F, Boriani G. Atrioventricular junction ablation in patients with atrial fibrillation treated with cardiac resynchronization therapy: positive impact on ventricular arrhythmias, implantable cardioverter-defibrillator therapies and hospitalizations. Eur J Heart Fail. 2018 Oct;20(10):1472-1481. doi: 10.1002/ejhf.1117. Epub 2017 Dec 18. PMID 29251799
- [Derived] Gasparini M, Anselme F, Clementy J, Santini M, Martinez-Ferrer J, De Santo T, Santi E, Schwab JO; ADVANCE CRT-D Investigators. BIVentricular versus right ventricular antitachycardia pacing to terminate ventricular tachyarrhythmias in patients receiving cardiac resynchronization therapy: the ADVANCE CRT-D Trial. Am Heart J. 2010 Jun;159(6):1116-1123.e2. doi: 10.1016/j.ahj.2010.02.007. PMID 20569728

RESULTS

PARTICIPANT FLOW:
Groups:
- Right Ventricle (RV): Anti Tachyarrhythmia Pacing (ATP) therapies are delivered in the right ventricle
- Biventricular (BiV): Anti Tachyarrhythmia Pacing (ATP) are delivered in both ventricles
Period: Overall Study
Arm/Group | Right Ventricle (RV) | Biventricular (BiV)
Started | 266 | 260
Completed | 266 | 260
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Right Ventricle (RV) | Biventricular (BiV) | Total
Number analyzed (Participants) | 266 | 260 | 526
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 95 | 189
  >=65 years | 172 | 165 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.2) | 66.8 (9.5) | 66.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 42 | 77
  Male | 231 | 218 | 449
Region of Enrollment [Number; unit: participants]
  Italy | 122 | 127 | 249
  France | 67 | 61 | 128
  Germany | 48 | 46 | 94
  Spain | 22 | 20 | 42
  Israel | 5 | 4 | 9
  Portugal | 1 | 1 | 2
  United Kingdom | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Anti Tachycardia Pacing (ATP) Therapy (Burst, 8 Pulses, 88 %, 1 Sequence) to Terminate All Types of Ventricular Tachycardia.
Description: Termination of Ventricular Tachycardia is calculated as percentage of successfully terminated episodes, adjusted for multiple events with GEE method. This technique yields an average therapy efficacy and 95% CI that is based on number of patients, number of episodes per patient, and magnitude of the correlation between responses within patients.
Time Frame: one year
Measure: Number; unit: Percent of VT episodes terminated
Arm/Group | Right Ventricle (RV) | Biventricular (BiV)
Number analyzed (Participants) | 260 | 266
Percent of VT episodes terminated | 64.7 | 68.2

2. Secondary Outcome: Compare Efficacy of the First BiV and RV ATP to Terminate FVT
Time Frame: one year
Reporting Status: Not Posted

3. Secondary Outcome: Compare Efficacy of the First BiV and RV ATP to Terminate Slow VT
Time Frame: one year
Reporting Status: Not Posted

4. Secondary Outcome: Compare Efficacy of BiV and RV ATP (All ATP Therapies) to Terminate Slow VT
Time Frame: one year
Reporting Status: Not Posted

5. Secondary Outcome: Determine the Rate of Both FVT and VT Episodes Which Are Accelerated or Degenerates Into VF
Time Frame: one year
Reporting Status: Not Posted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No